CLINICAL TRIAL: NCT04948021
Title: Interest of the Kleihauer in Patients With Decreased Active Fetal Movements
Acronym: MAF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: MAF
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Fetal Movement Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fetomaternal hemorrhage is the passage of fetal red blood cells through the placental barrier into the maternal blood. This phenomenon frequently occurs in the third trimester for small quantities of blood < 0.5 ml and is without fetal consequences in rhesus positive patients.

This hemorrhage can sometimes be more important and be the cause of fetal anemia or even fetal death in utero.

Diagnostic confirmation is biological and is performed using the Kleihauer test. It is based on the identification by the biologist of fetal cells circulating in the maternal blood by counting acid-fast fetal cells under the microscope. It is therefore a time-consuming examination with significant inter- and intra-observer variability.

The clinical sign most often reported in the literature, and the earliest sign that may suggest fetomaternal hemorrhage complicated by fetal anemia, is a decrease in active fetal movements. However, this is an aspecific sign and is one of the most common reasons for consultation in obstetric emergencies.

DETAILED DESCRIPTION:
There are other arguments in favor of complicated fetomaternal hemorrhage: The fetal heart rate is often altered in severe fetal anemia, with sinusoidal rhythm being pathognomonic but uncommon. A slightly oscillating rhythm or variable decelerations are also found.

On ultrasound, peak systolic middle cerebral artery velocity > 1.5 MoM correlates with fetal anemia early before the appearance of hydrops.

Some studies show that peak systolic middle cerebral artery velocity correlates better with neonatal hemoglobin than the Kleihauer test, for which no threshold has been found to predict an unfavorable outcome. Thus, even if the Kleihauer test is positive, the positive predictive value for fetal anemia is low. The detection of a small amount of fetomaternal hemorrhage by Kleihauer in the absence of evidence of anemia could even be deleterious, potentially leading to an excess of additional investigations and obstetrical interventions.

The interest of systematically performing the Kleihauer test to search for fetomaternal hemorrhage is uncertain at this time because of the development and the undeniable contribution of ultrasound. However, in France, it is still carried out in most maternity wards in the absence of recommendations for any decrease in active fetal movements.

Only one article has looked specifically at fetomaternal hemorrhage in a group of patients consulting for a decrease in active fetal movements, calling into question its interest.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age ≥ 18 years
* French speaking patients
* Consultation for decreased active fetal movements
* Singleton pregnancies
* Gestational age between 24 weeks of amenorrhea and 41 weeks of amenorrhea +5 days

Exclusion Criteria:

* Patients under guardianship or curatorship
* Patients deprived of liberty
* Patients under court protection
* Patients who object to the use of their data for this research
* Fetal or neonatal anemia of documented cause other than fetomaternal hemorrhage
* Consultation for metrorrhagia
* Consultation for Abdominal Trauma
* Consultation for external maneuver version

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be performed on data from patients referred for decreased active fetal movements between 01/01/2015 and 12/31/2020, approximately 1000 patients in total.
Sampling Method: Non-Probability Sample
Enrollment: 1683 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the diagnostic performance of each of the two tests: Kleihauer test / Doppler + fetal heart rate for the diagnosis of neonatal anemia (by cord blood sampling) among patients presenting with decreased active fetal movements. | Day 1
  Statistical performance of tests (sensitivity, specificity, negative/positive predictive value and positive/negative likelihood ratio)

SECONDARY OUTCOMES:
To evaluate the diagnostic performance of the middle cerebral artery Doppler + fetal heart rate pair in comparison with the Kleihauer test for the diagnosis of neonatal anemia. | Day 1
  Comparison of the diagnostic performance of the Kleihauer test and peak systolic middle cerebral artery velocity for neonatal anemia
To describe of obstetric outcomes for fetomaternal hemorrhage in patients consulting for decreased active fetal movements. | Day 1
  Adverse neonatal outcomes
To describe of obstetric outcomes for fetomaternal hemorrhage in patients consulting for decreased active fetal movements. | Day 1
  Adverse obstetrical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Inès BELAROUSSI, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France